CLINICAL TRIAL: NCT06848946
Title: Multicenter, Randomized, Double-masked, Parallel Group Trial to Evaluate the Safety and Efficacy of iDose® TR (Travoprost Intracameral Implant) in Conjunction With Cataract Surgery vs. Cataract Surgery Alone
Brief Title: Safety and Efficacy of iDose® TR With Cataract Surgery vs. Cataract Surgery Alone
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GLK-101-04
Record Dates: First submitted 2025-02-01; First posted 2025-02-27 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Glaucoma, Open-angle; Ocular Hypertension (OHT); Phacoemulsification Cataract Surgery
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- iDose TR (travoprost intracameral implant) 75 µg in conjunction with cataract surgery (Active Comparator): iDose TR (travoprost intracameral implant) 75 µg in conjunction with cataract surgery
  Interventions: Combination Product: iDose TR (travoprost intracameral implant) 75 µg in conjunction with cataract surgery
- Sham procedure in conjunction with cataract surgery (Sham Comparator): Sham procedure in conjunction with cataract surgery
  Interventions: Procedure: Sham procedure in conjunction with cataract surgery

INTERVENTIONS:
Combination Product: iDose TR (travoprost intracameral implant) 75 µg in conjunction with cataract surgery — iDose TR (travoprost intracameral implant) 75 µg in conjunction with cataract surgery
  Arms: iDose TR (travoprost intracameral implant) 75 µg in conjunction with cataract surgery
Procedure: Sham procedure in conjunction with cataract surgery — Sham procedure in conjunction with cataract surgery
  Arms: Sham procedure in conjunction with cataract surgery

SUMMARY:
This trial will evaluate the safety and IOP -lowering efficacy of administering an iDose TR (travoprost intracameral implant) in conjunction with cataract surgery compared to cataract surgery alone

DETAILED DESCRIPTION:
This is a Phase 4 randomized, double-masked, parallel group trial designed to evaluate the safety and IOP-lowering efficacy of administering iDose TR (travoprost intracameral implant 75 mcg) in conjunction with uncomplicated cataract surgery (phacoemulsification with a posterior chamber intraocular lens) compared to uncomplicated cataract surgery alone, in patients with open-angle glaucoma (OAG) or ocular hypertension (OHT).

ELIGIBILITY:
Inclusion Criteria:

* Cataract diagnosis: clinically significant age-related cataract eligible for phacoemulsification in the study eye.
* OAG or OHT diagnosis: either OAG (i.e. primary, pseudoexfoliation, or pigmentary glaucoma) or OHT in the study eye (i.e., eye to undergo cataract surgery)

Exclusion Criteria:

* Active corneal inflammation or edema.
* Retinal disorders not associated with glaucoma.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in mean diurnal IOP | 3 Months
  Mean diurnal IOP at the Month 3 Visit minus mean diurnal IOP at the Baseline Visit

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Chair — Glaukos Corporation
Locations (1):
- Glaukos Investigator Site, Kenosha, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No